CLINICAL TRIAL: NCT00584753
Title: Molecular Imaging of Breast Cancer With Breast PET/CT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Ramsey Badawi, Ph.D, Associate Professor, University of California, Davis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 200715040
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): Normal volunteers
  Interventions: Radiation: Positron emission tomography and computed tomography
- 2 (Active Comparator): Breast PET/CT scan
  Interventions: Radiation: Positron emission tomography and computed tomography
- 3 (Active Comparator): Whole body and breast PET/CT
  Interventions: Radiation: Positron emission tomography and computed tomography

INTERVENTIONS:
Radiation: Positron emission tomography and computed tomography — Positron emission tomography and computed tomography
  Other Names: Breast imaging
  Arms: 3
Radiation: Positron emission tomography and computed tomography — Positron emission tomography and computed tomography
  Other Names: Breast imaging
  Arms: 2
Radiation: Positron emission tomography and computed tomography — Positron emission tomography and computed tomography
  Other Names: Breast imaging
  Arms: 1

SUMMARY:
This study is a feasibility study to determine if a combined breast PET/CT scanner can image malignant functional activity while determining anatomical structure in the same clinical setting for patients with breast cancer. End-points of this study are whether women will accept the imaging position and timing, and whether functional properties of breast cancer can be imaged with this device. The secondary purpose of this study is to explore protocol parameters with a view to optimizing imaging performance whilst minimizing patient discomfort. Imaging results will be compared to histological samples to determine ground truth.

DETAILED DESCRIPTION:
PET is literally a molecular imaging modality. In monitoring the patient's response to a specific chemotherapeutic regime, baseline and subsequent PET/CT scans can be used to quantitatively determine the therapeutic effect of the regime, using the standard uptake value (SUV), a common metric in PET imaging. The breast PET/CT system will facilitate molecular imaging of breast cancer using a number of radiolabeled molecules, available both commercially (18-FDG) and from the research environment.

ELIGIBILITY:
Inclusion Criteria:

- Normal Adult Volunteers

* Female, at least 18 years of age
* Ability to lie motionless for up to 20 minutes

Patient Volunteers

* Female, at least 18 years of age
* Diagnostic findings from prior mammography highly suggestive of invasive breast carcinoma (BI-RADS category 5)
* Not pregnant or breast-feeding
* Ability to lie motionless for up to 20 minutes

Exclusion Criteria:

* Normal Adult Volunteers

  * Inability to understand the risks and benefits of the study

Patient Volunteers

* Recent breast biopsy
* Diagnostic findings from prior mammography highly suggestive of noninvasive ductal or lobular carcinoma
* Uncontrolled diabetes
* Diabetic and blood sugar level > 200 mg/dL
* Positive urine pregnancy test or currently breast-feeding
* Inability to understand the risks and benefits of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
End-points of this study are whether women will accept the imaging position and timing, and whether functional properties of breast cancer can be imaged with this device. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ramsey Badawi, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC David Medical Center, Sacramento, California, United States